CLINICAL TRIAL: NCT00873457
Title: Phase II Trial of Perifosine in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Perifosine in Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daphne Friedman (Other)
Collaborators: Keryx Biopharmaceuticals (Industry); Keryx / AOI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daphne Friedman, Medical Instructor, Medicine - Hematological Malignancies, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00015060
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: B-Cell Chronic Lymphocytic Leukemia; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perifosine (Experimental): Perifosine 50 mg twice a day for a total of six 28-day cycles.
  Interventions: Drug: perifosine

INTERVENTIONS:
Drug: perifosine — Perifosine 50 mg will be taken orally twice a day for a maximum of six 28-day cycles
  Other Names: D-21266

SUMMARY:
Perifosine inhibits the AKT pathway (a way cells communicate with each other). This pathway is felt to be important in the development of several types of cancers including chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). It is thought perifosine may be able to block this pathway and lead to an improvement in the CLL or SLL. The purpose of this trial is to see if perifosine is an effective treatment for relapsed or refractory CLL or SLL. Another purpose of this study is to look at the effect perifosine has on cells.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia and small B-cell lymphocytic lymphoma represent different manifestations of the same disease. CLL/SLL (hereafter denoted by CLL) is a clonal disorder of small B lymphocytes expressing a characteristic morphology and immunophenotype. The B cells express CD19, dim CD 20, dim CD 5, CD 23, CD 43, CD 79a, and weakly express surface immunoglobin. CLL can present asymptomatically in 25% of patients when diagnosed on a complete blood count. It also can present with diffuse painless lymphadenopathy and, in a smaller number of patients, B symptoms.

CLL is characterized by accumulation of circulating B cells predominantly in the G0 phase of the cell cycle. These cells are resistant to apoptosis. CLL has been found to have aberrant signaling in several pathways including NF-kB, Akt/PI3K, and JNK/STAT pathways. Akt is important in promoting CLL survival and viability, as seen in in vitro experiments where blocking its activity results in apoptosis. Thus an AKT inhibitor may lead to increased apoptosis and may have a role in the treatment of this disease.

Treatment options for CLL range from a watch and wait approach to high dose chemotherapy with stem cell support. Currently, there is no consensus on the best treatment regimen, since no treatment has been shown to improve survival in randomized prospective clinical trials. New approaches to treatment, especially those with lower toxicity rates, are needed.

Perifosine has been shown to inhibit or otherwise modify signaling through a number of different signal transduction pathways, including Akt, MAPK, and JNK. These pathways are involved in the development of cancers and resistance to chemotherapy. Perifosine is of particular interest, especially due to the difficulty in discovery of drugs that inhibit these pathways with minimal toxicity. The effect of perifosine on CLL cells has been tested in the laboratory and has been shown to be an active agent against primary CLL cells in vitro.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CLL or SLL based on iwCLL diagnostic criteria.
* Prior therapy for CLL (no limit on number of prior regimens).
* Patients requiring therapy, based on at least one of the iwCLL criteria.
* 18 years of age or older.
* Performance status ECOG 0, 1, or 2.
* An estimated or measured creatinine clearance ≥30 ml/min at study enrollment.
* AST, ALT, and total bilirubin ≤ 2.5 times the upper limit of normal, unless due to CLL/SLL.
* Female subject who is either post-menopausal or surgically sterilized or male or female subject willing to use an acceptable method of birth control for the duration of the study therapy and for 2 weeks after study therapy completion.

Exclusion Criteria:

* Female subject is pregnant or lactating.
* Patient has received other investigational drugs for this disease within 14 days of enrollment.
* Patient with known HIV prior to enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with another malignancy within the last three years (from documentation of remission) other than basal or squamous cell skin cancer or CIS of the cervix or early stage prostate cancer not requiring systemic treatment.
* Patients who underwent allogeneic stem cell transplant and have at least 2% donor cells engrafted will be excluded.
* Significant cardiac or vascular events within 6 months: acute MI, unstable angina, severe peripheral vascular disease (ischemic pain at rest class 3 or worse, non-healing ulcers/wounds, congestive heart failure (NHYA class ≥ 2), uncontrolled cardiac arrhythmias.
* Known severe hypersensitivity to perifosine or any component of the formulation.
* Life expectancy less than six months due to co-morbid illness
* Active autoimmune hemolytic anemia or immune thrombocytopenia, requiring current steroid therapy.
* De novo prolymphocytic leukemia (PLL) or PLL arising from CLL (≥ 55% prolymphocytes).
* Richter's transformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Friedman, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from Duke University Medical Center between 8/2009 and 7/2011
Pre-assignment Details: One patient was a screen failure and did not go on to participate in the study.
Period: Overall Study
Arm/Group | Perifosine
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Perifosine
Number analyzed (Participants) | 16
Age Continuous [Median (Full Range); unit: years] | 69.5 [62 to 87]
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Per International Workshop on Chronic Lymphocytic Leukemia, Complete Response (CR):normal CBC; absence of the following: clonal lymphocytes in blood and marrow, lymphadenopathy, hepatomegaly or splenomegaly, and constitutional symptoms; and bone marrow has <30% lymphocytes, is normocellular, and is without B-lymphoid nodules. Partial Response(PR): one of the following: decrease lymphadenopathy ≥ 50%; decrease of liver and/or spleen size ≥ 50%, any constitutional symptoms, Polymorphonuclear leukocytes ≥ 1,500/µl or a 50% improvement, or decrease of circulating clonal B lymphocytes ≥ 50% AND one of the following: Platelets ≥ 100,000/µl or a 50% improvement, Hemoglobin ≥ 11.0 g/dl or a 50% improvement, Bone marrow has ≥ 30% lymphocytes, or B-lymphoid nodules, or not done. Overall Response (OR)= CR+PR
Time Frame: after 3 months of treatment
Population: Patients who completed 3 months of therapy.
Measure: Number; unit: participants
Arm/Group | Perifosine
Number analyzed (Participants) | 8
participants | 1

2. Primary Outcome: Overall Response
Description: as for outcome 1
Time Frame: after 6 months of treatment
Population: Patients who completed 6 months of therapy
Measure: Number; unit: participants
Arm/Group | Perifosine
Number analyzed (Participants) | 1
participants | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the length of time between discontinuation of perifosine until death or 2 year's followup, whichever comes first.
Time Frame: up to a maximum of 2 years
Population: All treated patients
Measure: Median (Full Range); unit: Days
Arm/Group | Perifosine
Number analyzed (Participants) | 16
Days | 289.5 [19 to 730]

4. Secondary Outcome: Event-free Survival
Description: Event-free survival will be defined as the length of time between the discontinuation of study treatment and disease progression, next therapy, or death,whichever comes first, up to a maximum of 2 years.
Time Frame: up to a maximum of 2 years
Population: All treated patients
Measure: Median (Full Range); unit: Days
Arm/Group | Perifosine
Number analyzed (Participants) | 16
Days | 118 [19 to 350]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the initiation of study drug until 30 days after the last dose
Arm/Group | Perifosine
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perifosine (N=16)
Platelets (Investigations) | 1 (1)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Infection without febrile neutropenia (Infections and infestations) | 1 (1)
Edema: limb (General disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hemorrhage, GI (Gastrointestinal disorders) | 2 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 3 (3)
Infection - Other (Infections and infestations) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perifosine (N=16)
Platelets (Investigations) | 8 (8)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Infection - Other (Infections and infestations) | 3 (3)
Edema: limb (General disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 10 (10)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 4 (4)
Neutrophils / granulocytes (ANC / AGC) (Investigations) | 5 (7)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (14)
Insomnia (Psychiatric disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatology / Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hair Loss / Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus / itching (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes / flushes (Vascular disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Heartburn / dyspepsia (Gastrointestinal disorders) | 2 (2)
Mucositis / Stomatitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Taste Alteration (dysgeusia) (Nervous system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hemorrhage, pulmonary / upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema: Other (General disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Investigations) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (4)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4)
Mood Alteration - Agitation (Psychiatric disorders) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Ocular / Visual - Other (Eye disorders) | 1 (1)
Vision - blurred vision (Eye disorders) | 1 (1)
Vision - flashing lights / floaters (Eye disorders) | 1 (1)
Pain, Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Pain, Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (10)
Pain, Neurology (Nervous system disorders) | 3 (3)
Pain, Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Other (General disorders) | 2 (2)
Pain, Pulmonary / Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary / Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice changes / dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency / urgency (Renal and urinary disorders) | 1 (1)
Infection with unknown ANC - Ungual (nails) (Infections and infestations) | 1 (1)
Pain, chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Extremity-lower (gait / walking) (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. All patients were heavily pretreated and had aggressive disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes